CLINICAL TRIAL: NCT01744951
Title: Evaluate the Adoption-specific Prevention Treatment Program (ADAPT)
Brief Title: Adoption-specific Treatment Prevention Pilot Trial
Acronym: ADAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Center for Adoption Support and Education (Unknown)
Responsible Party: Principal Investigator, Dr. Jeanne Miranda, Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ADAPT-02; UCLA IRB/IRB# 12-001024 (Other Grant/Funding Number: Annie E Casey Foundation/212.0023)
Record Dates: First submitted 2012-11-28; First posted 2012-12-07 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Prevent Disorders in Children Adopted From Foster Care
Keywords: Adoption; Foster care; Substance abuse; Older children; Mental health
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADAPT (Experimental): ADAPT is a manualized intervention with eight treatment modules designed as an early intervention for children, ages 5-14, who are being adopted from foster care and their adoptive parent/s.
  Interventions: Behavioral: ADAPT
- Care as usual (No Intervention): Children, ages 5-14, and their adoptive parent/s will receive care as usual in the treatment setting.

INTERVENTIONS:
Behavioral: ADAPT — ADAPT consists of the following modules/sessions:
  Module 1: Trust, positive coping strategies, and behavior management; Module 2: Developmental understanding of adoption experience; Module 3: Substance abuse prevention; Module 4: Loss and grief issues about birth family and foster care; Module 5: Attachment/joining with adoptive family; Module 6: Search for identity/self -esteem; Module 7: Adoption and the outside world; Module 8: Trauma Treatment (if appropriate)
  Arms: ADAPT

SUMMARY:
This study seeks to pilot a manualized adoption-specific intervention aimed at providing a preventive intervention for families adopting children ages 5-14 years where family reunification has been terminated and the family is moving toward adoption or who have adopted children from foster care in the last three years. This work will fill a major gap in services to children and families and is developed to improve mental health and family functioning of children adopted from foster care, as well as decrease adoption disruptions. President Clinton's 1997 adoption initiative, The Adoption and Safe Families ACT (ASFA), along with subsequent Congressional initiatives, have provided incentives to States and subsidies for adopting older children with a resultant increase in rates of adoption from foster care from 26,000 in 1995 to 53,000 (stabilized annual rate) beginning in 2002. The mean age at adoption from foster care is now 6 years old. These older children have histories of physical and sexual abuse, neglect, and multiple placements, all factors that predict behavior problems over time. To address this gap in our knowledge of providing care for this vulnerable group, we have developed a manualized adoption-specific intervention for families adopting children from foster care. Because adoptive children generally enter homes with stable, well-functioning parents, interventions may be particularly effective in helping the children adjust and their parents learn to understand and manage children with difficult past histories.

The aim of this current pilot trial is to test this intervention designed to improve the outcomes for children adopted from foster care through a randomized trial. Our hypothesis is that this manualized adoption-specific intervention will be more effective than care as usual in improving child mental health and family functioning outcomes; specifically, families and children who have been randomized to the manualized adoption-specific intervention will show better outcomes on the post-treatment measures and the 3 month follow-up than on the pre-treatment measures than the care as usual families and children.

ELIGIBILITY:
Inclusion Criteria:

* Children being adopted from foster care, ages 5-14
* Children (within above age range) who have been adopted in the last three years
* Family reunification services have been terminated

Exclusion Criteria:

* Children with the following Diagnostic and Statistical Manual psychiatric disorders will be excluded from study participation: Pervasive Developmental Disorders (e.g. Asperger's, autism, mental retardation, or psychotic disorder as known to the parents
* Children will be excluded if the child has a major neurological disorder or a major medical illness that would interfere with participation in the study
* Children who pose a significant risk for dangerousness to self or others that makes participating inadvisable
* Children and/or parents who are non-English speaking and unable to complete treatment without a translator will not be included

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Parent Weekly Report | Participants will be followed for the duration of the therapeutic intervention, an expected average of 24 weeks.
  The Parent Weekly Report consists of two measures: Brief Problem Checklist (Chorpita et al., 2010 and Parent Daily Report (Chamberlain & Reid, 1987).

SECONDARY OUTCOMES:
Number of child participants whose internalizing and externalizing behaviors improve | 0 weeks, 24 weeks, 36 weeks
  Child participants' internalizing and externalizing behaviors will be measured at the three distinct times by using both child and parent measures: 1. Emotional Distress and Functioning:Children's Depression Inventory, Screen for Childhood Anxiety Related Emotional Disorders (SCARED),Child PTSD Symptom Scale (CPSS),Achenbach Child Behavior Checklists and Teacher Report Forms (CBCL),Children's Global Assessment Scale (CGAS) 2.Targeted Resilience Factors: Emotion Regulation Checklist (ER Checklist),Kidcope 3.Understanding of Adoption: Adoption Dynamics Questionnaire (ADQ),Children's Beliefs about Adoption Scale (CBAAS) 4.Family Environment and Parental Distress,Family Environment Scale (FES),Brief Symptom Inventory (BSI) 5.Attachment and Parenting: Inventory of Parent and Peer Attachment (IPPA) 6.Trauma Exposure: Modified Life Events Scale (LES) 7.Process Variables: Therapeutic Alliance Scale for Children (TASC),Working Alliance Inventory (WAI),Consumer Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Miranda, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - Children's Bureau of Southern California, Los Angeles, California
  - UCLA TIES for Familes, Los Angeles, California
  - UCLA TIES for Families South Bay, Torrance, California
  - Center for Adoption Support and Education, Burtonsville, Maryland
  - Children's Home Society North Carolina, Greensboro, North Carolina